CLINICAL TRIAL: NCT00908362
Title: Investigator Initiated, Placebo Controlled, Randomized Pilot Trial on the Influence of Fluticasone and Salmeterol on Airway Dendritic Cells (DCs) in Smokers With COPD Stage GOLD 0 or 1.
Brief Title: Impact of Fluticasone and Salmeterol on Airway Dendritic Cells (DCs) in Smokers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Rostock (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: University of Rostock, University of Rostock
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: LO-0003
Record Dates: First submitted 2009-05-20; First posted 2009-05-25 (Estimated); Last update posted 2010-01-13 (Estimated); Status verified 2009-05

CONDITIONS: Smoke-related Lung Diseases; Chronic Obstructive Pulmonary Disease
Keywords: Dendritic cells; Airway; Smoker; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Fluticasone; Fluticasone-Salmeterol Drug Combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Active Comparator): Inhalation of Fluticasone (via discus) twice daily for 28 days
  Interventions: Drug: fluticasone
- B (Active Comparator): Inhalation of Fluticasone and Salmeterol (via discus) twice daily for 28 days
  Interventions: Drug: fluticasone/salmeterol
- C (Placebo Comparator): Inhalation of Placebo (via discus) twice daily for 28 days.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: fluticasone — Participants inhale fluticasone (250 µg) via discus. Before and after this therapy, a bronchoalveolar lavage is performed.
  Arms: A
Drug: fluticasone/salmeterol — Participants inhale fluticasone/salmeterol (250/50µg) via discus. Before and after this therapy, a bronchoalveolar lavage is performed.
  Arms: B
Drug: placebo — Participants inhale placebo twice daily via discus. Before and after this therapy, a bronchoalveolar lavage is performed.
  Arms: C

SUMMARY:
Airway dendritic cells (DCs) play a key role in smoke-related lung diseases. In this study, the researchers investigate the effects of fluticasone and salmeterol on human airway DCs in smokers. The researchers hypothesize that fluticasone and salmeterol impact on the number and the characteristics of airway DCs in smokers.

ELIGIBILITY:
Inclusion Criteria:

* Men aged 30 - 60 years
* At least 15 years of smoking
* Current smoker, at least 10 cigarettes per day

Exclusion Criteria:

* Any acute or chronic disease (except COPD oder hypertension)
* Any regular medication (except drugs against hypertension)
* FEV1 < 80% predicted
* Oxygen saturation < 90%
* Acute infections of the lower respiratory tract in the last 7 days before the first day of the study

Ages: 30 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2009-05; Primary Completion 2009-10 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
The number and the CCR7 expression of DCs in bronchoalveolar lavage fluid before and after therapy with fluticasone or fluticasone/salmeterol, as compared to placebo. | 2 time points (A and B). Time point A: day 0 (directly before the inhalation therapy). Time point B: day 29 (directly after the inhalation therapy).

SECONDARY OUTCOMES:
The expression of other surface molecules on DCs in bronchoalveolar lavage fluid before and after therapy with fluticasone or fluticasone/salmeterol, as compared to placebo. | 2 time points (A and B). Time point A: day 0 (directly before the inhalation therapy). Time point B: day 29 (directly after the inhalation therapy).

CONTACTS AND LOCATIONS:
Locations (1):
- Dep. of Pneumology, University of Rostock, Rostock, Mecklenburg-Vorpommern, Germany

REFERENCES:
- [Background] Bratke K, Klug M, Bier A, Julius P, Kuepper M, Virchow JC, Lommatzsch M. Function-associated surface molecules on airway dendritic cells in cigarette smokers. Am J Respir Cell Mol Biol. 2008 Jun;38(6):655-60. doi: 10.1165/rcmb.2007-0400OC. Epub 2008 Jan 18. PMID 18203971
- [Derived] Lommatzsch M, Kraeft U, Troebs L, Garbe K, Bier A, Stoll P, Klammt S, Kuepper M, Bratke K, Virchow JC. Fluticasone impact on airway dendritic cells in smokers: a randomized controlled trial. Respir Res. 2013 Oct 29;14(1):114. doi: 10.1186/1465-9921-14-114. PMID 24168756